CLINICAL TRIAL: NCT01856491
Title: RELIANCE 4-FRONT™ Passive Fixation Defibrillation Lead Post Market Clinical Follow-Up (PMCF) Study
Brief Title: Safety and Performance Study of the RELIANCE 4-Front Passive Fixation Lead
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1868
Record Dates: First submitted 2013-05-15; First posted 2013-05-17 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Tachycardia; Ventricular Fibrillation; Ventricular Flutter
Keywords: RELIANCE 4-FRONT; Implantable Cardioverter Defibrillator (ICD); Cardiac Resynchronization Therapy - Defibrillator (CRT-D)
MeSH Terms: conditions — Tachycardia; Ventricular Fibrillation; Ventricular Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- RELIANCE 4-FRONT™ Passive Fixation (Other): Single arm, all patients will be implanted with the RELIANCE 4-FRONT™ Passive Fixation lead
  Interventions: Device: RELIANCE 4-FRONT™ Passive Fixation lead implantation

INTERVENTIONS:
Device: RELIANCE 4-FRONT™ Passive Fixation lead implantation — Implantation of transvenous defibrillation lead with passive fixation mechanism.

SUMMARY:
The objective of this study is to gather data to establish the chronic safety, performance and effectiveness of the RELIANCE 4-FRONT™ Passive Fixation Defibrillation Leads.

DETAILED DESCRIPTION:
The RELIANCE 4-FRONT Passive Fixation Defibrillation Lead Post Market Clinical Follow-Up Study is a prospective, non-randomized, multi-center, single-group, post market clinical study to establish the chronic safety, performance and effectiveness of the RELIANCE 4-FRONT passive fixation defibrillation leads.

A total of 167 patients (including 10 % attrition) are required to evaluate the Primary Endpoint.

Up to 10 Investigational centers located in Europe and Israel. Lead-related Complication-Free Rate (CFR) from Implant through 3 Months Post-Implant.

Lead-related complications associated with the RELIANCE 4-FRONT passive fixation lead will count toward this endpoint.

Lead-related Complication-Free Rate from 3 Months through 15 Months Post-Implant.

Lead-related complications associated with the RELIANCE 4-FRONT passive fixation lead will count toward this endpoint.

* Lead-related Complication-Free Rate from 3 Months through 24 Months Post-Implant
* Pacing Threshold at 0.5 ms pulse width at 3 Months Post-Implant
* Sensed Amplitude at 3 Months Post-Implant
* Pacing Impedance at 3 Months Post-Implant All endpoints will be assessed for the RELIANCE 4-FRONT passive fixation lead.

Clinic visits will occur at:

* Enrollment Visit (no later than 30 days prior to implant procedure)
* Implant Procedure (Day 0; all future follow ups based on this date)
* Pre-Discharge Clinic Visit (3 - 72 hours post-implant)
* One Month Clinic Visit (30±7 days)
* 3 Month Clinic Visit (91 ± 21 days)
* 6 Month Clinic Visit (180 ± 30 days)
* 12 Month Clinic Visit (365 ± 45 days)
* 18 Month Clinic Visit (545± 45 days)
* 24 Month Clinic Visit (730 ± 45 days) The study will be considered completed after all subjects have completed the 24 Month follow-up and study completion is anticipated in 2015. Primary endpoint completion is anticipated after all subjects have completed the 3 Month follow-up visit. All study required visits will be completed during clinic visits.

Hypotheses testing in the RELIANCE 4-FRONT passive fixation PMCF Study will use standard statistical methodology as specified more in detail in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Willing and capable of providing informed consent
* Has an indication for implantation of a single or dual chamber ICD or CRT-D system in their respective geography
* Subjects planned to be implanted with the RELIANCE 4-FRONT Passive Fixation Lead
* Willing and capable of participating in all testing/ visits associated with this clinical study at an approved clinical study center and at the intervals defined by this protocol
* Age 18 or above, or of legal age to give informed consent specific to state and national law

Exclusion Criteria:

* Known or suspected sensitivity to Dexamethasone Acetate (DXA)
* Mechanical tricuspid heart valve
* Subject is enrolled in any other concurrent study without prior written approval from Boston Scientific (BSC), with the exception of local mandatory governmental registries and observational studies/registries that are not in conflict and do not affect the following:
* Schedule of procedures for the RELIANCE 4-Front Study (i.e. should not cause additional or missed visits);
* RELIANCE 4-Front Study outcome (i.e. involve medications that could affect the heart rate of the subject);
* Conduct of the RELIANCE 4-Front Study per Good Clinical Practice (GCP)/ International Organization for Standardization (ISO) 14155:2011/ 21 CFR 812/ local regulations
* Currently on the active heart transplant list
* Documented life expectancy of less than 12 months
* Women of childbearing potential who are or might be pregnant at the time of study enrollment (method of assessment upon physician discretion)
* Currently requiring chronic dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2015-11-02 (Actual); Study Completion 2017-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia Bongiorni, MD, Principal Investigator — University Hospital Pisa, Italy
Locations (11):
- German Heart Center, Berlin, Germany
- Israel (3):
  - Meir Medical Center, Kfar Saba
  - Beilinson Medical Center, Petah Tikva
  - Sheba Medical Center, Tel Litwinsky
- Italy (7):
  - Fondazione di Ricerca e Cura 'Giovanni Paolo II, Campobasso
  - Ospedale Alessandro Manzoni, Lecco
  - Clinica Mediterranea, Naples
  - Ospedale Buon Consiglio, Naples
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Osp. Civile S. Maria Delle Grazie, Pozzuoli
  - Ospedale San Pietro Fatebenefratelli, Rome

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RELIANCE 4-FRONT™ Passive Fixation
Started | 167
Completed | 152
Not Completed | 15

BASELINE CHARACTERISTICS:
Arm/Group | RELIANCE 4-FRONT™ Passive Fixation
Number analyzed (Participants) | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.90 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 134
Race (NIH/OMB) [Count of Participants; unit: Participants] — Patient demographic data has been collected during the enrollment visit. No study-specific collection was conducted prior to consent.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 166
    More than one race | 0
    Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Complication Free Rate
Description: Lead-related Complication-Free Rate (CFR) from Implant through 3 Months Post-Implant.
Time Frame: 3-months
Population: 167 have been enrolled. 165 were included in the analysis because for 2 patients the leads have not been implanted
Measure: Number (95% Confidence Interval); unit: percentage of patients without event
Arm/Group | RELIANCE 4-FRONT™ Passive Fixation
Number analyzed (Participants) | 165
percentage of patients without event | 97.5 [94.4 to 100]

2. Secondary Outcome: Complication Free Rate
Description: Lead-related Complication-Free Rate from 3 Months through 15 Months Post-Implant.
Time Frame: 3 months through 15 months post implant
Population: Subjects were eligible for the secondary endpoint analysis if their date of last follow-up was ≥92 days post-implant procedure.
Measure: Number (95% Confidence Interval); unit: percentage of patients without events
Arm/Group | RELIANCE 4-FRONT™ Passive Fixation
Number analyzed (Participants) | 158
percentage of patients without events | 99.4 [95 to 100]

3. Other Pre Specified Outcome: Pacing Threshold at 0.5 ms Pulse Width
Description: Pacing Threshold at 0.5 ms pulse width at 3 Months Post-Implant. During the RELIANCE 4-FRONT PASSIVE fixation PMCF Study pacing threshold measurements are collected from RELIANCE 4-FRONT PASSIVE fixation leads in the standard manual fashion. At least 3 cardiac cycles at a given voltage level shall be obtained before stepping down to the next voltage level. A count of two non-capture beats is required at a given voltage level to declare a loss of capture (LOC) for any of these tests. The threshold is defined as one voltage level above the level where two non-captured beats are observed. Threshold tests must be taken with a pulse width of 0.5 ms.
Time Frame: 3 Months Post-Implant
Population: 167 have been enrolled. 138 were included in the analysis because we have the lead measurements for those number of patients collected .
Measure: Mean (Standard Deviation); unit: Volt
Arm/Group | RELIANCE 4-FRONT™ Passive Fixation
Number analyzed (Participants) | 138
Volt | 0.48 (0.59)

4. Other Pre Specified Outcome: Complication Free Rate
Description: Lead-related Complication-Free Rate from 3 Months through 24 Months Post-Implant
Time Frame: 3 months through 24 months post implant
Measure: Number (95% Confidence Interval); unit: percentage of patients without events
Arm/Group | RELIANCE 4-FRONT™ Passive Fixation
Number analyzed (Participants) | 158
percentage of patients without events | 99.4 [95 to 100]

5. Other Pre Specified Outcome: Sensed Amplitude
Description: Lead performance evaluations of the Reliance 4-FRONT PASSIVE fixation lead have been conducted in accordance with the Physician's Lead Manual. Measurements should fall within the recommended values as mentioned below:
  Signal Type Amplitude Pacing Threshold Impedance Pacing/Sensing ≥ 5mV ≤1.5 V 300-1200 Ω Defibrillation ≥ 1mV N/A 20-125 Ω The required data from the implant procedure for the study lead is measured with a pacing system analyzer (PSA) to verify adequate signals. Electrical performance of the lead was verified before attaching the lead to the Pulse Generator (PG). After the PG has been implanted evaluation of the study lead using the PG has been performed. Lead measurements were required unless the testing is prohibited by a subject's condition (subject has no intrinsic rhythm). In case the measurements are variable (e.g. in patients with atrial fibrillation), the most reproducible value has been collected.
Time Frame: 3 Months Post-Implant
Population: 167 patients were enrolled. From 141 patients we could collected the sensed amplitude at 3 months
Measure: Mean (Standard Deviation); unit: mVolt
Arm/Group | RELIANCE 4-FRONT™ Passive Fixation
Number analyzed (Participants) | 141
mVolt | 18.5 (5.7)

6. Other Pre Specified Outcome: Pacing Impedance
Description: as for outcome 5
Time Frame: 3 Months Post-Implant
Population: 167 patients have been enrolled. For 150 patients we were able to collect the 3 month pacing impedance
Measure: Mean (Standard Deviation); unit: Ohm
Arm/Group | RELIANCE 4-FRONT™ Passive Fixation
Number analyzed (Participants) | 150
Ohm | 474 (106)

ADVERSE EVENTS:
Time Frame: 3-month follow-up data
Arm/Group | RELIANCE 4-FRONT™ Passive Fixation
All-Cause Mortality (participants affected / at risk) | 4/167
Serious Adverse Events (participants affected / at risk) | 84/167
Other Adverse Events (participants affected / at risk) | 55/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RELIANCE 4-FRONT™ Passive Fixation (N=167)
Inappropriate tachy therapy - SVT (Cardiac disorders) | 1 (1)
Erosion (Skin and subcutaneous tissue disorders) | 1 (1)
Infection (> 30 days post-implant) (Infections and infestations) | 3 (3)
Psychological effect due to device therapy (Psychiatric disorders) | 1 (2)
Post-surgical wound discomfort (Skin and subcutaneous tissue disorders) | 1 (1)
Post-surgical infection (<= 30 days post-implant) (Infections and infestations) | 2 (2)
Chest pain (Cardiac disorders) | 1 (1)
Hematoma - Pocket (<=30 days post-implant) (Skin and subcutaneous tissue disorders) | 4 (4)
Conductor coil fracture - RA (General disorders) | 1 (1)
Elevated threshold - RV (General disorders) | 2 (2)
Dislodgment - Unable to capture - LV (General disorders) | 1 (1)
Pneumothorax - Procedure (Injury, poisoning and procedural complications) | 2 (3)
Ventricular fibrillation (VF) (Cardiac disorders) | 3 (3)
Ventricular tachycardia (VT) (Cardiac disorders) | 3 (6)
Atrial flutter (Cardiac disorders) | 3 (3)
Other SVT (AVRT, AVNRT, EAT etc.) (Cardiac disorders) | 1 (1)
Chest pain - Heart failure (Cardiac disorders) | 3 (3)
Dyspnea - Heart failure (Cardiac disorders) | 8 (11)
Peripheral edema - Heart failure (Cardiac disorders) | 1 (1)
Pulmonary edema - Heart failure (Cardiac disorders) | 4 (6)
Heart failure symptoms - Unspecified (Cardiac disorders) | 6 (8)
Multiple heart failure symptoms (Cardiac disorders) | 4 (5)
Multi-system failure - Heart failure (Cardiac disorders) | 5 (5)
Hypotension (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
RELATED TO ISCHEMIA (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 6 (6)
Coronary Artery Disease (Vascular disorders) | 2 (2)
Coronary artery disease (Vascular disorders) | 1 (1)
Peripheral vascular disease (Vascular disorders) | 3 (4)
Intermittent claudication (Vascular disorders) | 1 (1)
Mitral regurgitation (Cardiac disorders) | 1 (2)
Syncope (Cardiac disorders) | 3 (4)
Dizziness (Cardiac disorders) | 2 (3)
Chest pain - Ischemic (Cardiac disorders) | 1 (2)
Chest pain - Other (Cardiac disorders) | 6 (7)
Fatigue (General disorders) | 1 (1)
Cerebrovascular accident (CVA) (Vascular disorders) | 6 (6)
Pulmonary embolism (PE) (Vascular disorders) | 1 (1)
Intracardiac thrombus (Vascular disorders) | 1 (1)
Hematoma - Unrelated to procedure or device (General disorders) | 1 (1)
Death (General disorders) | 4 (4)
Systemic infection (Infections and infestations) | 2 (2)
Fever (General disorders) | 2 (2)
Physical trauma (Injury, poisoning and procedural complications) | 2 (2)
Abnormal laboratory values (Blood and lymphatic system disorders) | 3 (4)
Hematological (Blood and lymphatic system disorders) | 5 (7)
Neurological (Nervous system disorders) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 10 (11)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 9 (13)
Genitourinary (Renal and urinary disorders) | 7 (14)
Renal (Renal and urinary disorders) | 7 (9)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (2)
Integumentary (Skin and subcutaneous tissue disorders) | 1 (1)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 2 (2)
Endocrine (Endocrine disorders) | 2 (2)
Multi-system failure (General disorders) | 1 (1)
sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RELIANCE 4-FRONT™ Passive Fixation (N=167)
Not yet classified (General disorders) | 3 (4)
Inappropriate tachy therapy - SVT (Cardiac disorders) | 4 (5)
Inappropriate tachy therapy - Other (Cardiac disorders) | 1 (1)
Post-surgical wound discomfort (Surgical and medical procedures) | 1 (1)
Inadvertent VT/VF (Cardiac disorders) | 2 (2)
Hematoma - Pocket (<=30 days post-implant) (Injury, poisoning and procedural complications) | 2 (2)
Elevated threshold - RA (Cardiac disorders) | 1 (1)
Elevated threshold - RV (Cardiac disorders) | 1 (1)
Coronary venous dissection (Vascular disorders) | 1 (1)
Ventricular fibrillation (VF) (Cardiac disorders) | 2 (2)
Ventricular tachycardia (VT) (Cardiac disorders) | 1 (1)
Atrial fibrillation (AF) (Cardiac disorders) | 4 (5)
Other SVT (AVRT, AVNRT, EAT etc.) (Cardiac disorders) | 3 (3)
Syncope - Heart failure (Cardiac disorders) | 1 (1)
Chest pain - Heart failure (Cardiac disorders) | 1 (1)
Dyspnea - Heart failure (Cardiac disorders) | 7 (8)
Multiple heart failure symptoms (Cardiac disorders) | 1 (1)
Hypertension - Heart failure (Cardiac disorders) | 1 (1)
Chest pain - Ischemic (Cardiac disorders) | 1 (1)
Chest pain - Other (Cardiac disorders) | 7 (7)
Palpitations (Cardiac disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
Hemorrhage (Surgical and medical procedures) | 1 (1)
Physical trauma (General disorders) | 6 (6)
Hematological (Blood and lymphatic system disorders) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 5 (10)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Genitourinary (Renal and urinary disorders) | 4 (5)
Renal (Renal and urinary disorders) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 6 (12)
Psychological (Psychiatric disorders) | 1 (1)
Integumentary (Skin and subcutaneous tissue disorders) | 3 (5)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 10 (12)
Endocrine (Endocrine disorders) | 2 (2)
Cancer (General disorders) | 2 (4)
medication side effect (General disorders) | 1 (1)
pain in device pocket (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Sample size is rather small and the power of the study is only 80%

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less